CLINICAL TRIAL: NCT06058806
Title: Effects of Multimodal Physical Therapy on Pain, Disability, H-reflex, and Diffusion Tensor Imaging Parameters in Patients With Lumbosacral Radiculopathy
Brief Title: Effects of Multimodal Physical Therapy in Patients With Lumbosacral Radiculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Badr Hassanein, Mr, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MBH18
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Lumbosacral Radiculopathy
Keywords: Lumbosacral Radiculopathy; Lumbar disc herniation
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multimodal Physical Therapy (Experimental): Patients in this group will receive Multimodal Physical Therapy program consisting of electrophysical agents, manual therapy interventions, and core stability exercises.
  Interventions: Other: Multimodal Physical Therapy

INTERVENTIONS:
Other: Multimodal Physical Therapy — Multimodal Physical Therapy program consisting of electrophysical agents, manual therapy interventions, and core stability exercises
  Other Names: Physical Therapy; Physiotherapy

SUMMARY:
Purposes of the study

To investigate the effect of Multimodal Physical Therapy on pain, daiablility H-reflex, and Diffusion Tensor Imaging (DTI) Parameters in Patients With Lumbosacral Radiculopathy.

DETAILED DESCRIPTION:
Participants will receive Multimodal Physical Therapy program consisting of electrophysical agents, manual therapy interventions, and core stability exercises. Patients will receive the intervention for six weeks. Outcomes will be assessed at baseline and post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* chronic (≥ 3 months) unilateral Lumbosacral Radiculopathy (LSR)
* The LSR is due to paracentral L4-L5 or L5-S1 Lumbar disc herniation
* The LSR is confirmed radiologically by MRI
* The LSR is confirmed clinically by history and physical examination
* The LSR is confirmed neurophysiological by soleus H-reflex assessment
* Body mass Index less than 30
* 20-45 years of age

Exclusion Criteria:

* systematic disease
* Bilateral symptoms
* Lumbar spinal stenosis
* previous surgery
* Steroid injection
* Spinal fracture
* Lumbar spinal stenosis
* Spinal deformity
* Spinal fracture
* Radiological evidence of bilateral nerve root encroachmen
* Evidence of H-reflex amplitude or latency affection on asymptomatic side

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Pain | Change from Baseline pain at 6 weaks
  Visual analog scale (VAS)
Disability | Change from Baseline Disability at 6 weaks
  Roland-Morris Disability Questionnaire (RMDQ)
Soleus H-reflex amplitude | Change from Baseline Soleus H-reflex amplitude at 6 weaks
  by EMG unit
Soleus H-reflex side-to-side amplitude (H/H) ratio | Change from Baseline Soleus H/H ratio at 6 weaks
  by EMG unit
Fractional anisotropy (FA) of the compressed nerve root | Change from Baseline Fractional anisotropy (FA) ratio at 6 weaks
  by MRI examination
Apparent diffusion coefficient (ADC) of the compressed nerve root | Change from Baseline Apparent diffusion coefficient (ADC) at 6 weaks
  by MRI examination

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Cairo University, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided